CLINICAL TRIAL: NCT04465071
Title: Patient Satisfaction,Dry Symptoms in Patients Cataract Surgery in NHS Patients Treated With Prophylactic Preservative-free Lubricant Eye Drops (AEONTM Repair, and AEONTM Protect Plus): A Randomized, Prospective, Controlled Study.
Brief Title: Lubricating Eye Drops After Routine Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: City, University of London (Other); King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 276400
Record Dates: First submitted 2020-02-21; First posted 2020-07-09 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Dry Eye; Cataract
MeSH Terms: conditions — Dry Eye Syndromes; Cataract | interventions — Lubricant Eye Drops

STUDY DESIGN:
Intervention Model Description: To assess the use of additional lubricant eye-drops for 6 weeks following uncomplicated, routine cataract sur-gery to improve patient satisfaction and symptoms of dry eye in an NHS (public health care) setting, compared to no additional lubricating eye drops
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Treatment (No Intervention): Post-Cataract surgery standard treatment of Maxidex 0.1% QDS for 4 weeks, and Chloramphenicol drops QDS for 2 weeks
- Standard Treatment plus lubricating drops (Other): Lubricant eye-drops (0.3% cross linked sodium hyaluronate, AEONTM Protect Plus and phosphate-free, preservative-free lubricant eye drops containing 0.15% Sodium Hyaluronate with vita-mins A and E (AEONTM Repair) for 6 weeks post-Cataract surgery, in addition to the standard treatment of Maxidex 0.1% QDS for 4 weeks, and Chloramphenicol drops QDS for 2 weeks
  Interventions: Drug: AEONTM Repair and AEONTM Protect Plus lubricating eye drops

INTERVENTIONS:
Drug: AEONTM Repair and AEONTM Protect Plus lubricating eye drops — AEONTM Repair and AEONTM Protect Plus lubricating eye drops
  Arms: Standard Treatment plus lubricating drops

SUMMARY:
Patient satisfaction and dry symptoms in patients undergoing routine uncomplicated cataract surgery in NHS patients treated with prophylactic phosphate-free, preservative-free lubricant eye drops (0.3% cross linked sodium hyaluronate, AEONTM Protect Plus and0.15% Sodium Hyalu-ronate with vitamins A and E, AEONTM Repair): A randomized, prospective, controlled study.

DETAILED DESCRIPTION:
The aim of this study is to investigate the routine use of such lubricating drops in a randomized, prospective methodology in patients undergoing uncomplicated cataract surgery in the NHS setting. As these drops are provided with the intraocular lens, if found to be of benefit in reducing dry eye problems such a study might provide evidence for the universal implementa-tion of post-operative ocular lubricant drops

ELIGIBILITY:
Inclusion Criteria:

1. Bilateral or unilateral cataracts requiring surgical intervention
2. Age over 18 years
3. Able to understand informed consent and the objectives of the trial
4. Not pregnant, not breast feeding
5. No previous eye surgery

Exclusion Criteria:

1. age-related macula degeneration
2. glaucoma
3. previous retinal vascular disorders
4. previous retinal detachment or tear
5. any neuro-ophthalmological condition
6. any inherited retinal disorder or pathology
7. previous strabismus surgery or record of amblyopia
8. previous TIA, CVA or other vaso-occlusive disease
9. already enrolled in another study
10. already on prescribed lubricating drops

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
CATPROM 5 patient satisfaction score | Baseline, 2 week follow up and 2 month follow up. Measure scores at three times points to assess for any change
  Quality of life patient satisfaction questionnaire
EQ5D3L patient satisfaction score | Baseline, 2 week follow up and 2 month follow up. Measure scores at three times points to assess for any change
  Quality of life patient satisfaction questionnaire
Dry Eye Symptoms | Baseline, 2 week follow up and 2 month follow up. Measure scores at three times points to assess for any change
  Patient questionnaire SPEED II score (Maximum 28, Minimum 0)

SECONDARY OUTCOMES:
Visual Acuity | 2 week follow up and 2 month follow up
  Logmar Visual Acuity
Cornea and Conjunctival Staining | 2 week follow up and 2 month follow up
  Oxford Scale (Maximum 5, minimum 0)
Schirmer 1 Test | 2 week follow up and 2 month follow up
  Schirmer 1 Test (Normal >10 mm)
Tear Break up time | 2 week follow up and 2 month follow up
  Non-invasive tear breakup time (normal >10 seconds)
Inferior tear meniscus | 2 week follow up and 2 month follow up
  Inferior tear meniscus
Corneal Incision site and size | 2 week follow up and 2 month follow up
  Corneal Incision site and size

CONTACTS AND LOCATIONS:
Locations (1):
- Guys' and St.Thomas' Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No